CLINICAL TRIAL: NCT01658631
Title: Evaluation of Nexfin During Induction of General Anesthesia and in Intensive Care During a Passive Legs Raising Test
Brief Title: Evaluation of Nexfin During Anesthesia and in Intensive Care (NexfinEval)
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/42; 2010-A00881-38 (Other: ANSM)
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anesthesia: Arterial pressure measurement using Nexfin (a noninvasive finger cuff system) during the induction of anesthesia
  Interventions: Device: arterial pressure measurement (Nexfin, a noninvasive finger cuff system)
- Intensive Care Unit patients: Arterial pressure measurement using Nexfin (a noninvasive finger cuff system) during a passive legs raising test
  Interventions: Device: arterial pressure measurement (Nexfin, a noninvasive finger cuff system)

INTERVENTIONS:
Device: arterial pressure measurement (Nexfin, a noninvasive finger cuff system)

SUMMARY:
The purpose of this study is to compare the non invasive measurement of arterial pressure (Nexfin monitor)with the invasive measurement of arterial pressure (radial artery catheter)

* during induction of general anesthesia,
* during a leg raising test in the Intensive Care Unit

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* ASA II, III or IV
* weight between 40 and 180 kg; BMI < 35
* normal Allen's test and/or hand Doppler examination.

Exclusion Criteria:

* cardiac arrhythmias,
* history of vascular surgery or vascular implant in the upper limb
* Raynaud disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major surgery with the need for an invasive blood pressure measurement and ICU patients requiring a passive legs raising test
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Arterial pressure measurement | Blood pressure will be followed for the duration of induction of anesthesia, an expected average of 20 minutes, or for the passive legs raising test, an expected average of 20 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Mutualiste Montsouris, Paris
  - Hopital Foch, Suresnes

REFERENCES:
- [Derived] Weiss E, Gayat E, Dumans-Nizard V, Le Guen M, Fischler M. Use of the Nexfin device to detect acute arterial pressure variations during anaesthesia induction. Br J Anaesth. 2014 Jul;113(1):52-60. doi: 10.1093/bja/aeu055. Epub 2014 Apr 25. PMID 24771806